CLINICAL TRIAL: NCT04081090
Title: Structured Cognitive Therapy to Improve Neurocognitive Dysfunction in Older Intensive Care Unit Sepsis Survivors
Brief Title: Clinical Translational Science Institute (CTSI) Brain HQ Modules vs. Active Controls for Elderly Survivors of ICU
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Delay due to COVID. Lost funding.
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Rahul Nanchal, Associate Professor of Medicine, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 32542
Record Dates: First submitted 2019-04-30; First posted 2019-09-09 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Neurocognitive Disorders
MeSH Terms: conditions — Neurocognitive Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brain HQ adaptive Cognitive Therapy Modules (Experimental): Brain HQ licensed modules that adapt to each individuals unique strengths and weaknesses to address deficits and improve neuroplasticity.
  Interventions: Behavioral: Brain HQ Cognitive Modules
- Brain HQ Active Control Modules (Active Comparator): Participants in this arm will complete puzzles such as crossword puzzles, Sudoku, etc.
  Interventions: Behavioral: Brain HQ Cognitive Modules

INTERVENTIONS:
Behavioral: Brain HQ Cognitive Modules — Online personalized cognitive therapy modules to address and improve neuroplasticity.

SUMMARY:
The purpose of this project is to test whether an online cognitive rehabilitation program or online thinking exercises helps improve memory and thinking in elderly patients who survive a severe infection.

DETAILED DESCRIPTION:
Currently, over 50% of patients are estimated to develop an Alzheimer's like disease following their hospitalization. This means they might have trouble remembering simple things or doing simple tasks. This can make returning to normal life difficult. This project will test whether online thinking exercises can help speed up patient's recovery.

ELIGIBILITY:
Inclusion Criteria:

1. Admitted to the Intensive Care Unit (ICU) at Froedtert Memorial Lutheran Hospital (FMLH)
2. Diagnosis of Sepsis
3. Age 65 years or older
4. Required mechanical ventilation or vasopressor therapy while in the ICU
5. Had delirium while in the ICU

Exclusion Criteria:

1. Non-English Speaking
2. Severe Dementia that would interfere with the ability to participate in the study activities
3. Prior or current structural neurological injury that would confound study results
4. Inability to communicate for any reason
5. Current chemotherapy or radiation treatment
6. Recent history of substance abuse
7. Life expectancy < 6 months
8. Planned discharge to long term acute care facility or nursing home
9. Lack reliable access to the internet either through a computer or smart device

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-08-26 (Actual)

PRIMARY OUTCOMES:
Tailored Online Cognitive Rehabilitation | 3 months
  Older survivors of sepsis will demonstrate > 80% adherence to a tailored cognitive rehabilitation program
Adherence to Online Intervention Modules | 3 months
  In recruited survivors of sepsis investigator will measure adherence to a facilitated structured neurocognitive rehabilitation program (administered as one-hour sessions, three days per week for 3 months) via a computer or smart device/phone.

SECONDARY OUTCOMES:
Improvement in Neurocognitive Function part 1 | 6 months
  A structured cognitive rehabilitation program will significantly improve neurocognitive function in older survivors of sepsis as measured by Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) 40 - 160 scale measuring Immediate Memory, Visuospatial/Constructional, Language, Attention and Delayed Memory , Delis-Kaplan Executive Function System (D-KEFS) Trail Making Test.
Improvement in Neurocognitive Function part 2 | 6 months
  A structured cognitive rehabilitation program will significantly improve neurocognitive function in older survivors of sepsis as measured by Delis-Kaplan Executive Function System (D-KEFS) Trail Making Test and Symbol-Digit Modality Test measuring the duration it takes to complete the test.
Measure Differences in Cognitive Performance | 6 months
  Investigators will measure differences in cognitive performance at 3 and 6 months using the above mentioned tests in participants with active neurocognitive rehabilitation intervention as compared to controls. Consistent with the National Academy of Medicine recommendations the control group will receive an active intervention. This will include mind stimulating games such as Brain HQ crossword puzzles and Sudoku modules measuring the ability to complete and duration.

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Nanchal, MD, MS, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Memorial Lutheran Hospital, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual data collected as part of this project.

REFERENCES:
- [Background] Ely EW, Shintani A, Truman B, Speroff T, Gordon SM, Harrell FE Jr, Inouye SK, Bernard GR, Dittus RS. Delirium as a predictor of mortality in mechanically ventilated patients in the intensive care unit. JAMA. 2004 Apr 14;291(14):1753-62. doi: 10.1001/jama.291.14.1753. PMID 15082703
- [Background] Pandharipande P, Cotton BA, Shintani A, Thompson J, Pun BT, Morris JA Jr, Dittus R, Ely EW. Prevalence and risk factors for development of delirium in surgical and trauma intensive care unit patients. J Trauma. 2008 Jul;65(1):34-41. doi: 10.1097/TA.0b013e31814b2c4d. PMID 18580517
- [Background] McPherson JA, Wagner CE, Boehm LM, Hall JD, Johnson DC, Miller LR, Burns KM, Thompson JL, Shintani AK, Ely EW, Pandharipande PP. Delirium in the cardiovascular ICU: exploring modifiable risk factors. Crit Care Med. 2013 Feb;41(2):405-13. doi: 10.1097/CCM.0b013e31826ab49b. PMID 23263581
- [Background] McNicoll L, Pisani MA, Zhang Y, Ely EW, Siegel MD, Inouye SK. Delirium in the intensive care unit: occurrence and clinical course in older patients. J Am Geriatr Soc. 2003 May;51(5):591-8. doi: 10.1034/j.1600-0579.2003.00201.x. PMID 12752832
- [Background] Pisani MA, Murphy TE, Van Ness PH, Araujo KL, Inouye SK. Characteristics associated with delirium in older patients in a medical intensive care unit. Arch Intern Med. 2007 Aug 13-27;167(15):1629-34. doi: 10.1001/archinte.167.15.1629. PMID 17698685
- [Background] Tsuruta R, Oda Y, Shintani A, Nunomiya S, Hashimoto S, Nakagawa T, Oida Y, Miyazaki D, Yabe S; Japanese Epidemiology of Delirium in ICUs (JEDI) Study Investigators. Delirium and coma evaluated in mechanically ventilated patients in the intensive care unit in Japan: a multi-institutional prospective observational study. J Crit Care. 2014 Jun;29(3):472.e1-5. doi: 10.1016/j.jcrc.2014.01.021. Epub 2014 Feb 3. PMID 24602999
- [Background] Lat I, McMillian W, Taylor S, Janzen JM, Papadopoulos S, Korth L, Ehtisham A, Nold J, Agarwal S, Azocar R, Burke P. The impact of delirium on clinical outcomes in mechanically ventilated surgical and trauma patients. Crit Care Med. 2009 Jun;37(6):1898-905. doi: 10.1097/CCM.0b013e31819ffe38. PMID 19384221
- [Background] Hsieh SJ, Soto GJ, Hope AA, Ponea A, Gong MN. The association between acute respiratory distress syndrome, delirium, and in-hospital mortality in intensive care unit patients. Am J Respir Crit Care Med. 2015 Jan 1;191(1):71-8. doi: 10.1164/rccm.201409-1690OC. PMID 25393331
- [Background] Milbrandt EB, Deppen S, Harrison PL, Shintani AK, Speroff T, Stiles RA, Truman B, Bernard GR, Dittus RS, Ely EW. Costs associated with delirium in mechanically ventilated patients. Crit Care Med. 2004 Apr;32(4):955-62. doi: 10.1097/01.ccm.0000119429.16055.92. PMID 15071384
- [Background] Almeida IC, Soares M, Bozza FA, Shinotsuka CR, Bujokas R, Souza-Dantas VC, Ely EW, Salluh JI. The impact of acute brain dysfunction in the outcomes of mechanically ventilated cancer patients. PLoS One. 2014 Jan 22;9(1):e85332. doi: 10.1371/journal.pone.0085332. eCollection 2014. PMID 24465538
- [Background] Gunther ML, Morandi A, Krauskopf E, Pandharipande P, Girard TD, Jackson JC, Thompson J, Shintani AK, Geevarghese S, Miller RR 3rd, Canonico A, Merkle K, Cannistraci CJ, Rogers BP, Gatenby JC, Heckers S, Gore JC, Hopkins RO, Ely EW; VISIONS Investigation, VISualizing Icu SurvivOrs Neuroradiological Sequelae. The association between brain volumes, delirium duration, and cognitive outcomes in intensive care unit survivors: the VISIONS cohort magnetic resonance imaging study*. Crit Care Med. 2012 Jul;40(7):2022-32. doi: 10.1097/CCM.0b013e318250acc0. PMID 22710202
- [Background] Girard TD, Jackson JC, Pandharipande PP, Pun BT, Thompson JL, Shintani AK, Gordon SM, Canonico AE, Dittus RS, Bernard GR, Ely EW. Delirium as a predictor of long-term cognitive impairment in survivors of critical illness. Crit Care Med. 2010 Jul;38(7):1513-20. doi: 10.1097/CCM.0b013e3181e47be1. PMID 20473145
- [Background] Girard TD, Thompson JL, Pandharipande PP, Brummel NE, Jackson JC, Patel MB, Hughes CG, Chandrasekhar R, Pun BT, Boehm LM, Elstad MR, Goodman RB, Bernard GR, Dittus RS, Ely EW. Clinical phenotypes of delirium during critical illness and severity of subsequent long-term cognitive impairment: a prospective cohort study. Lancet Respir Med. 2018 Mar;6(3):213-222. doi: 10.1016/S2213-2600(18)30062-6. PMID 29508705
- [Background] Wolters AE, van Dijk D, Pasma W, Cremer OL, Looije MF, de Lange DW, Veldhuijzen DS, Slooter AJ. Long-term outcome of delirium during intensive care unit stay in survivors of critical illness: a prospective cohort study. Crit Care. 2014 Jun 18;18(3):R125. doi: 10.1186/cc13929. PMID 24942154
- [Background] van den Boogaard M, Schoonhoven L, Evers AW, van der Hoeven JG, van Achterberg T, Pickkers P. Delirium in critically ill patients: impact on long-term health-related quality of life and cognitive functioning. Crit Care Med. 2012 Jan;40(1):112-8. doi: 10.1097/CCM.0b013e31822e9fc9. PMID 21926597
- [Background] Jackson JC, Girard TD, Gordon SM, Thompson JL, Shintani AK, Thomason JW, Pun BT, Canonico AE, Dunn JG, Bernard GR, Dittus RS, Ely EW. Long-term cognitive and psychological outcomes in the awakening and breathing controlled trial. Am J Respir Crit Care Med. 2010 Jul 15;182(2):183-91. doi: 10.1164/rccm.200903-0442OC. Epub 2010 Mar 18. PMID 20299535
- [Background] Needham DM, Dinglas VD, Morris PE, Jackson JC, Hough CL, Mendez-Tellez PA, Wozniak AW, Colantuoni E, Ely EW, Rice TW, Hopkins RO; NIH NHLBI ARDS Network. Physical and cognitive performance of patients with acute lung injury 1 year after initial trophic versus full enteral feeding. EDEN trial follow-up. Am J Respir Crit Care Med. 2013 Sep 1;188(5):567-76. doi: 10.1164/rccm.201304-0651OC. PMID 23805899
- [Background] Iwashyna TJ, Ely EW, Smith DM, Langa KM. Long-term cognitive impairment and functional disability among survivors of severe sepsis. JAMA. 2010 Oct 27;304(16):1787-94. doi: 10.1001/jama.2010.1553. PMID 20978258
- [Background] Iwashyna TJ, Cooke CR, Wunsch H, Kahn JM. Population burden of long-term survivorship after severe sepsis in older Americans. J Am Geriatr Soc. 2012 Jun;60(6):1070-7. doi: 10.1111/j.1532-5415.2012.03989.x. Epub 2012 May 29. PMID 22642542
- [Background] Morandi A, Rogers BP, Gunther ML, Merkle K, Pandharipande P, Girard TD, Jackson JC, Thompson J, Shintani AK, Geevarghese S, Miller RR 3rd, Canonico A, Cannistraci CJ, Gore JC, Ely EW, Hopkins RO; VISIONS Investigation, VISualizing Icu SurvivOrs Neuroradiological Sequelae. The relationship between delirium duration, white matter integrity, and cognitive impairment in intensive care unit survivors as determined by diffusion tensor imaging: the VISIONS prospective cohort magnetic resonance imaging study*. Crit Care Med. 2012 Jul;40(7):2182-9. doi: 10.1097/CCM.0b013e318250acdc. PMID 22584766
- [Background] Fong TG, Davis D, Growdon ME, Albuquerque A, Inouye SK. The interface between delirium and dementia in elderly adults. Lancet Neurol. 2015 Aug;14(8):823-832. doi: 10.1016/S1474-4422(15)00101-5. Epub 2015 Jun 29. PMID 26139023
- [Background] van der Kooi AW, Slooter AJ, van Het Klooster MA, Leijten FS. EEG in delirium: Increased spectral variability and decreased complexity. Clin Neurophysiol. 2014 Oct;125(10):2137-9. doi: 10.1016/j.clinph.2014.02.010. Epub 2014 Feb 23. No abstract available. PMID 24631011
- [Background] van Dellen E, van der Kooi AW, Numan T, Koek HL, Klijn FA, Buijsrogge MP, Stam CJ, Slooter AJ. Decreased functional connectivity and disturbed directionality of information flow in the electroencephalography of intensive care unit patients with delirium after cardiac surgery. Anesthesiology. 2014 Aug;121(2):328-35. doi: 10.1097/ALN.0000000000000329. PMID 24901239
- [Background] Choi SH, Lee H, Chung TS, Park KM, Jung YC, Kim SI, Kim JJ. Neural network functional connectivity during and after an episode of delirium. Am J Psychiatry. 2012 May;169(5):498-507. doi: 10.1176/appi.ajp.2012.11060976. PMID 22549209
- [Background] Reade MC, Eastwood GM, Bellomo R, Bailey M, Bersten A, Cheung B, Davies A, Delaney A, Ghosh A, van Haren F, Harley N, Knight D, McGuiness S, Mulder J, O'Donoghue S, Simpson N, Young P; DahLIA Investigators; Australian and New Zealand Intensive Care Society Clinical Trials Group. Effect of Dexmedetomidine Added to Standard Care on Ventilator-Free Time in Patients With Agitated Delirium: A Randomized Clinical Trial. JAMA. 2016 Apr 12;315(14):1460-8. doi: 10.1001/jama.2016.2707. PMID 26975647
- [Background] Girard TD, Kress JP, Fuchs BD, Thomason JW, Schweickert WD, Pun BT, Taichman DB, Dunn JG, Pohlman AS, Kinniry PA, Jackson JC, Canonico AE, Light RW, Shintani AK, Thompson JL, Gordon SM, Hall JB, Dittus RS, Bernard GR, Ely EW. Efficacy and safety of a paired sedation and ventilator weaning protocol for mechanically ventilated patients in intensive care (Awakening and Breathing Controlled trial): a randomised controlled trial. Lancet. 2008 Jan 12;371(9607):126-34. doi: 10.1016/S0140-6736(08)60105-1. PMID 18191684
- [Background] Schweickert WD, Pohlman MC, Pohlman AS, Nigos C, Pawlik AJ, Esbrook CL, Spears L, Miller M, Franczyk M, Deprizio D, Schmidt GA, Bowman A, Barr R, McCallister KE, Hall JB, Kress JP. Early physical and occupational therapy in mechanically ventilated, critically ill patients: a randomised controlled trial. Lancet. 2009 May 30;373(9678):1874-82. doi: 10.1016/S0140-6736(09)60658-9. Epub 2009 May 14. PMID 19446324
- [Background] Balas MC, Vasilevskis EE, Olsen KM, Schmid KK, Shostrom V, Cohen MZ, Peitz G, Gannon DE, Sisson J, Sullivan J, Stothert JC, Lazure J, Nuss SL, Jawa RS, Freihaut F, Ely EW, Burke WJ. Effectiveness and safety of the awakening and breathing coordination, delirium monitoring/management, and early exercise/mobility bundle. Crit Care Med. 2014 May;42(5):1024-36. doi: 10.1097/CCM.0000000000000129. PMID 24394627
- [Background] Skrobik Y, Ahern S, Leblanc M, Marquis F, Awissi DK, Kavanagh BP. Protocolized intensive care unit management of analgesia, sedation, and delirium improves analgesia and subsyndromal delirium rates. Anesth Analg. 2010 Aug;111(2):451-63. doi: 10.1213/ANE.0b013e3181d7e1b8. Epub 2010 Apr 7. PMID 20375300
- [Background] Dale CR, Kannas DA, Fan VS, Daniel SL, Deem S, Yanez ND 3rd, Hough CL, Dellit TH, Treggiari MM. Improved analgesia, sedation, and delirium protocol associated with decreased duration of delirium and mechanical ventilation. Ann Am Thorac Soc. 2014 Mar;11(3):367-74. doi: 10.1513/AnnalsATS.201306-210OC. PMID 24597599
- [Background] Bounds M, Kram S, Speroni KG, Brice K, Luschinski MA, Harte S, Daniel MG. Effect of ABCDE Bundle Implementation on Prevalence of Delirium in Intensive Care Unit Patients. Am J Crit Care. 2016 Nov;25(6):535-544. doi: 10.4037/ajcc2016209. PMID 27802955
- [Background] Page VJ, Ely EW, Gates S, Zhao XB, Alce T, Shintani A, Jackson J, Perkins GD, McAuley DF. Effect of intravenous haloperidol on the duration of delirium and coma in critically ill patients (Hope-ICU): a randomised, double-blind, placebo-controlled trial. Lancet Respir Med. 2013 Sep;1(7):515-23. doi: 10.1016/S2213-2600(13)70166-8. Epub 2013 Aug 21. PMID 24461612
- [Background] Trogrlic Z, van der Jagt M, Bakker J, Balas MC, Ely EW, van der Voort PH, Ista E. A systematic review of implementation strategies for assessment, prevention, and management of ICU delirium and their effect on clinical outcomes. Crit Care. 2015 Apr 9;19(1):157. doi: 10.1186/s13054-015-0886-9. PMID 25888230
- [Background] Buonomano DV, Merzenich MM. Cortical plasticity: from synapses to maps. Annu Rev Neurosci. 1998;21:149-86. doi: 10.1146/annurev.neuro.21.1.149. PMID 9530495
- [Background] Merzenich MM, Van Vleet TM, Nahum M. Brain plasticity-based therapeutics. Front Hum Neurosci. 2014 Jun 27;8:385. doi: 10.3389/fnhum.2014.00385. eCollection 2014. PMID 25018719
- [Background] Strenziok M, Parasuraman R, Clarke E, Cisler DS, Thompson JC, Greenwood PM. Neurocognitive enhancement in older adults: comparison of three cognitive training tasks to test a hypothesis of training transfer in brain connectivity. Neuroimage. 2014 Jan 15;85 Pt 3:1027-39. doi: 10.1016/j.neuroimage.2013.07.069. Epub 2013 Aug 6. PMID 23933474
- [Background] Zaal IJ, Devlin JW, Peelen LM, Slooter AJ. A systematic review of risk factors for delirium in the ICU. Crit Care Med. 2015 Jan;43(1):40-7. doi: 10.1097/CCM.0000000000000625. PMID 25251759
- [Background] Aldemir M, Ozen S, Kara IH, Sir A, Bac B. Predisposing factors for delirium in the surgical intensive care unit. Crit Care. 2001 Oct;5(5):265-70. doi: 10.1186/cc1044. Epub 2001 Sep 6. PMID 11737901
- [Background] Dubois MJ, Bergeron N, Dumont M, Dial S, Skrobik Y. Delirium in an intensive care unit: a study of risk factors. Intensive Care Med. 2001 Aug;27(8):1297-304. doi: 10.1007/s001340101017. PMID 11511942
- [Background] Lin SM, Huang CD, Liu CY, Lin HC, Wang CH, Huang PY, Fang YF, Shieh MH, Kuo HP. Risk factors for the development of early-onset delirium and the subsequent clinical outcome in mechanically ventilated patients. J Crit Care. 2008 Sep;23(3):372-9. doi: 10.1016/j.jcrc.2006.09.001. Epub 2007 Jan 31. PMID 18725043
- [Background] Ouimet S, Kavanagh BP, Gottfried SB, Skrobik Y. Incidence, risk factors and consequences of ICU delirium. Intensive Care Med. 2007 Jan;33(1):66-73. doi: 10.1007/s00134-006-0399-8. Epub 2006 Nov 11. PMID 17102966
- [Background] Robinson TN, Raeburn CD, Tran ZV, Angles EM, Brenner LA, Moss M. Postoperative delirium in the elderly: risk factors and outcomes. Ann Surg. 2009 Jan;249(1):173-8. doi: 10.1097/SLA.0b013e31818e4776. PMID 19106695
- [Background] Van Rompaey B, Elseviers MM, Schuurmans MJ, Shortridge-Baggett LM, Truijen S, Bossaert L. Risk factors for delirium in intensive care patients: a prospective cohort study. Crit Care. 2009;13(3):R77. doi: 10.1186/cc7892. Epub 2009 May 20. PMID 19457226
- [Background] van den Boogaard M, Pickkers P, Slooter AJ, Kuiper MA, Spronk PE, van der Voort PH, van der Hoeven JG, Donders R, van Achterberg T, Schoonhoven L. Development and validation of PRE-DELIRIC (PREdiction of DELIRium in ICu patients) delirium prediction model for intensive care patients: observational multicentre study. BMJ. 2012 Feb 9;344:e420. doi: 10.1136/bmj.e420. PMID 22323509
- [Background] Zaal IJ, Spruyt CF, Peelen LM, van Eijk MM, Wientjes R, Schneider MM, Kesecioglu J, Slooter AJ. Intensive care unit environment may affect the course of delirium. Intensive Care Med. 2013 Mar;39(3):481-8. doi: 10.1007/s00134-012-2726-6. Epub 2012 Oct 24. PMID 23093246
- [Background] Girard TD, Ware LB, Bernard GR, Pandharipande PP, Thompson JL, Shintani AK, Jackson JC, Dittus RS, Ely EW. Associations of markers of inflammation and coagulation with delirium during critical illness. Intensive Care Med. 2012 Dec;38(12):1965-73. doi: 10.1007/s00134-012-2678-x. Epub 2012 Aug 18. PMID 22903241
- [Background] Ohtake PJ, Lee AC, Scott JC, Hinman RS, Ali NA, Hinkson CR, Needham DM, Shutter L, Smith-Gabai H, Spires MC, Thiele A, Wiencek C, Smith JM. Physical Impairments Associated With Post-Intensive Care Syndrome: Systematic Review Based on the World Health Organization's International Classification of Functioning, Disability and Health Framework. Phys Ther. 2018 Aug 1;98(8):631-645. doi: 10.1093/ptj/pzy059. PMID 29961847
- [Background] Doiron KA, Hoffmann TC, Beller EM. Early intervention (mobilization or active exercise) for critically ill adults in the intensive care unit. Cochrane Database Syst Rev. 2018 Mar 27;3(3):CD010754. doi: 10.1002/14651858.CD010754.pub2. PMID 29582429
- [Background] Fleischmann C, Scherag A, Adhikari NK, Hartog CS, Tsaganos T, Schlattmann P, Angus DC, Reinhart K; International Forum of Acute Care Trialists. Assessment of Global Incidence and Mortality of Hospital-treated Sepsis. Current Estimates and Limitations. Am J Respir Crit Care Med. 2016 Feb 1;193(3):259-72. doi: 10.1164/rccm.201504-0781OC. PMID 26414292